CLINICAL TRIAL: NCT06842966
Title: A Prospective Multicenter Randomized Double-blind Placebo-controlled Study in Parallel Groups to Evaluate the Efficacy, Safety, and Tolerability of the Drug 4-MUST, Tablets, 128 mg Administered at Various Doses in Patients With Chronic Cholecystitis and Biliary Dyskinesia
Brief Title: Efficacy, Safety, and Tolerability of 4-MUST Tablets in Chronic Cholecystitis and Biliary Dyskinesia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Valenta Pharm JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GIB-02-03-2024
Record Dates: First submitted 2025-02-17; First posted 2025-02-24 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Chronic Cholecystitis; Biliary Dyskinesia
MeSH Terms: conditions — Biliary Dyskinesia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 4-MUST, 128 mg (Experimental): Patients will receive 1 tablet of the drug 4-MUST (128 mg of trimebutine 4-methylumbelliferyl sulfate) and 2 placebo tablets three times a day.
  Interventions: Drug: 4-MUST; Drug: Placebo
- 4-MUST, 256 mg (Experimental): Patients will receive 2 tablets of the drug 4-MUST (256 mg of trimebutine 4-methylumbelliferyl sulfate) and 1 placebo tablet three times a day.
  Interventions: Drug: 4-MUST; Drug: Placebo
- 4-MUST, 384 mg (Experimental): Patients will receive 3 tablets of the drug 4-MUST (384 mg of trimebutine 4-methylumbelliferyl sulfate) three times a day.
  Interventions: Drug: 4-MUST
- Placebo (Placebo Comparator): Patients will receive 3 placebo tablets three times a day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 4-MUST — 128 mg of trimebutine 4-methylumbelliferyl sulfate tablet.
  Other Names: trimebutine 4-methylumbelliferyl sulfate
  Arms: 4-MUST, 128 mg; 4-MUST, 256 mg; 4-MUST, 384 mg
Drug: Placebo — Placebo tablet.
  Arms: 4-MUST, 128 mg; 4-MUST, 256 mg; Placebo

SUMMARY:
This study aims to evaluate the efficacy, safety, and tolerability of the drug 4-MUST at various doses compared to placebo in patients with chronic cholecystitis and biliary dyskinesia

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18-70 years.
2. Presence of established gastrointestinal diseases: Chronic cholecystitis (K81.1); Dyskinesia of the bile duct or gallbladder (K82.8).
3. Presence of pain/discomfort in the upper abdomen combined with at least one of the following symptoms: Heartburn; Belching; Nausea; Abdominal bloating; Borborygmi (stomach rumbling); Flatulence; Constipation; Diarrhea.
4. Maximum severity of pain/discomfort in the upper abdomen over the past week is 40 mm or more on the VAS (Visual Analog Scale).
5. Severity of gastrointestinal symptoms according to the GSRS (Gastrointestinal Symptom Rating Scale) questionnaire is at least 30 points.
6. Women who are either sexually abstinent or using effective contraception methods (e.g. intrauterine devices, contraceptive patches, long-acting injectable contraceptives, or double barrier methods) for at least 8 weeks before and 3 weeks after the end of the study, with a confirmed negative pregnancy test, as well as women with documented infertility or non-childbearing status (e.g. hysterectomy, tubal ligation, infertility or menopause for more than 1 year) or men using barrier contraceptives throughout the study and for 3 weeks after its completion, or men unable to conceive (documented conditions: vasectomy, infertility).
7. Signed and dated informed consent from.

Non-inclusion Criteria:

1. Peptic ulcer disease, duodenal ulcer, erosive GERD.
2. Toxic megacolon.
3. Paralytic ileus.
4. Gilbert's syndrome.
5. Abdominal adhesion disease.
6. Blood in stool, unexplained weight loss, fever, anemia.
7. Inflammatory and erosive gastrointestinal diseases.
8. Irritable bowel syndrome, non-specific ulcerative colitis, Crohn's disease.
9. Oncological diseases of the gastrointestinal tract (including past diagnoses).
10. History of gastrointestinal surgical procedures, including but not limited to endoscopic papillotomy and cholecystectomy, exept for appendectomy.
11. Use of prohibited therapy medications within 3 days prior to randomization.
12. History of mental illnesses.
13. Chronic heart failure IIb-III stages and/or III-IV functional classes according to NYHA, angina pectoris III-IV functional classes.
14. Chronic kidney disease stage IIIa-V (according to NKF/KDOQI, 2006).
15. Established diagnosis of liver failure, including in history and/or changes in liver enzyme activity: Increase in AST, ALT, ALP and/or γ-GTP more than 3 times above the upper limit of normal; Increase in total bilirubin more than 2 times above the upper limit of normal or development of jaundice.
16. HIV, syphilis, viral hepatitis B or C, including in history.
17. Lactose intolerance, lactase deficiency, and glucose-galactose malabsorption syndrome.
18. Liver cirrhosis.
19. Hypersensitivity to the active ingridient or any of the excipients of the drug 4-MUST.
20. Severe, decompensated or unstable somatic diseases (any diseases or conditions that threaten the patient's life or worsen their prognosis and make it impossible for the patient to participate in clinical research).
21. Diabetes mellitus in a state of subcompensation and decompensation.
22. Systemic connective tissue diseases.
23. Autoimmune diseases.
24. Need for surgical and/or endovascular treatment and/or necessity for hemodialysis procedures.
25. Epilepsy or seizures of unclear etiology, including in history.
26. Alcoholism, substance abuse or drug addiction, including in history.
27. Uncorrected electrolyte disturbances.
28. History of surgery within 6 month prior to screening.
29. Women during pregnancy or lactation; women planning to become pregnant within the next 6 months.
30. Patients who require prohibited concomitant therapy within this study framework.
31. Participation in another clinical trial within the last 3 months prior to the screening visit date.
32. Lack of willingness to cooperate from the patient's side.
33. Other conditions that, in the investigator's judgement, may preclude the patient's participation in the study.

Exclusion Criteria:

1. Incorrect enrollment of a patient in the study (failure to meet inclusion/exclusion criteria at the time of randomization).
2. Ineffectiveness of therapy. The therapy will be deemed ineffective if there is no clinical improvement by visit 3 (15±1 days of therapy) - persistence or increase in the severity of pain/discomfort in the upper abdomen on the VAS compared to baseline. If excluded, the patient will be assigned alternative treatment at the discretion of the investigator.
3. Patient non-compliance (a compliant patient is defined as one who has taken at least 202 and no more than 303 tablets).
4. Requirement for prohibited concomitant therapy.
5. If the investigator judges that comtinued participation in the study would harm the patient.
6. Pregnancy or the need for breastfeeding in the patient.
7. Gross violation by the patient of the study protocol procedures outlined in the patient information sheet (PIS).
8. Withdrawal of informed consent (patient's unwillingness to continue participation in the study).
9. Loss of contact with the patient (inability to reach the patient via mobile and home phone (if applicable), as well as through a contact person; there must be at least three documented attempts to contact the patient).
10. Emergence during the study of any diseases or conditions that worsen the patient's prognosis, making it impossible for the patient to continue participating in this clinical trial.
11. Any other reasons, including administrative issues, that in the investigator's judgement may interfere with subject's ability to comlete the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Average reduction in the severity of pain/discomfort in the upper abdomen on the VAS by day 29 compared to baseline | Day 29 ± 1
  Visual analogue scale (VAS) from 0 to 100 mm, where 0 is "no pain", and 100 is "the worst pain one can imagine"

SECONDARY OUTCOMES:
Change in the total score of gastrointestinal symptom severity according to the GSRS questionnaire on days 8, 15, 22, and 29 compared to baseline | Day 8 ± 1, 15 ± 1, 22 ± 1, and 29 ± 1
  The Gastrointestinal Symptom Rating Scale (GSRS) is a self-administered questionnaire designed to assess gastrointestinal symptoms and their severity. It consists of 15 items categorized into five domains: Abdominal pain (including stomach pain and nausea), Reflux (heartburn and acid reflux), Indigestion (bloating, burping, and flatulence), Constipation (hard stools and incomplete evacuation), Diarrhea (loose stools and urgency). Respondents rate their symptoms on a 7-point Likert scale, where 1 indicates no discomfort and 7 indicates very severe discomfort.
Response rate to therapy (proportion of patients in the group showing a reduction in pain/discomfort in the upper abdomen on the VAS by more than 30%) by day 29 compared to baseline | Day 29 ± 1
  Visual analogue scale (VAS) from 0 to 100 mm, where 0 is "no pain", and 100 is "the worst pain one can imagine"
Response rate to therapy (proportion of patients in the group showing a reduction in pain/discomfort in the upper abdomen on the VAS by 50% or more) by day 29 compared to baseline | Day 29 ± 1
  Visual analogue scale (VAS) from 0 to 100 mm, where 0 is "no pain", and 100 is "the worst pain one can imagine"
Change in manifestations of dyspeptic disorders according to the GSRS questionnaire scores on days 8, 15, 22, and 29 compared to baseline | Day 8 ± 1, 15 ± 1, 22 ± 1, and 29 ± 1
  The Gastrointestinal Symptom Rating Scale (GSRS) is a self-administered questionnaire designed to assess gastrointestinal symptoms and their severity. It consists of 15 items categorized into five domains: Abdominal pain (including stomach pain and nausea), Reflux (heartburn and acid reflux), Indigestion (bloating, burping, and flatulence), Constipation (hard stools and incomplete evacuation), Diarrhea (loose stools and urgency). Respondents rate their symptoms on a 7-point Likert scale, where 1 indicates no discomfort and 7 indicates very severe discomfort.
Change in quality of life based on the total score from the SF-36 questionnaire by day 29 compared to baseline | Day 29 ± 1
  SF-36 (Short Form 36 Health Survey) is a self-reported questionnaire. It consists of 36 items that cover eight health domains: Physical functioning, Role limitations due to physical health, Role limitations due to emotional problems, Bodily pain, General health perceptions, Vitality (energy and fatigue), Social functioning, Mental health. SF-36 produces a profile of scores for each domain, which can be summarized into two main components: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). Scores range from 0 to 100, where lower scores indicate greater disability and higher scores indicate better health.
Average reduction in pain/discomfort severity in the upper abdomen on the VAS by days 8, 15, and 22 compared to baseline | Day 8 ± 1, 15 ± 1, 22 ± 1, and 29 ± 1
  Visual analogue scale (VAS) from 0 to 100 mm, where 0 is "no pain", and 100 is "the worst pain one can imagine"
Safety and Tolerability: adverse event (AE) rate | From the date of screening (and signing informed consent form) to the end of the study or to an early termination visit, whichever came first, assessed up to day 36 ± 2 for each participant
  Frequency of adverse events (AEs) or serious AEs (SAEs)
Safety and Tolerability: adverse event (AE) number | From the date of screening (and signing informed consent form) to the end of the study or to an early termination visit, whichever came first, assessed up to day 36 ± 2 for each participant
  Number of adverse events (AEs) or serious AEs (SAEs)
Safety and Tolerability: AEs associated with the study drug | From the date of screening (and signing informed consent form) to the end of the study or to an early termination visit, whichever came first, assessed up to day 36 ± 2 for each participant
  Number and frequency of AEs associated with the study drug
Safety and Tolerability: SAEs associated with the study drug | From the date of screening (and signing informed consent form) to the end of the study or to an early termination visit, whichever came first, assessed up to day 36 ± 2 for each participant
  Number and frequency of SAEs associated with the study drug
Safety and Tolerability: treatment discontinuation | From the date of screening (and signing informed consent form) to the end of the study or to an early termination visit, whichever came first, assessed up to day 36 ± 2 for each participant
  Percentage of patients who discontinued treatment due to the occurrence of AEs/SAEs
Safety and Tolerability: vital signs - systolic blood pressure (SBP) | Screening, day 1, day 8 ± 1, day 15 ± 1, day 22 ± 1, day 29 ± 1
  SBP, mmHg
Safety and Tolerability: vital signs - diastolic blood pressure (DBP) | Screening, day 1, day 8 ± 1, day 15 ± 1, day 22 ± 1, day 29 ± 1
  DBP, mmHg
Safety and Tolerability: vital signs - respiratory rate (RR) | Screening, day 1, day 8 ± 1, day 15 ± 1, day 22 ± 1, day 29 ± 1
  RR, breaths per minute
Safety and Tolerability: vital signs - heart rate (HR) | Screening, day 1, day 8 ± 1, day 15 ± 1, day 22 ± 1, day 29 ± 1
  HR, beats per minute
Safety and Tolerability: vital signs - body temperature | Screening, day 1, day 8 ± 1, day 15 ± 1, day 22 ± 1, day 29 ± 1
  Body temperature, Celsius scale
Physical examination results: cardiovascular system | Screening, day 1, day 8 ± 1, day 15 ± 1, day 22 ± 1, day 29 ± 1
  An assessment of the condition of the cardiovascular system on physical examination (normal condition or list of abnormal conditions, if any)
Physical examination results: respiratory system | Screening, day 1, day 8 ± 1, day 15 ± 1, day 22 ± 1, day 29 ± 1
  An assessment of the condition of the respiratory system on physical examination (normal condition or list of abnormal conditions, if any)(normal condition or list of abnormal conditions, if any)
Physical examination results: digestive tract | Screening, day 1, day 8 ± 1, day 15 ± 1, day 22 ± 1, day 29 ± 1
  An assessment of the condition of the digestive tract on physical examination (normal condition or list of abnormal conditions, if any)
Physical examination results: endocrine system | Screening, day 1, day 8 ± 1, day 15 ± 1, day 22 ± 1, day 29 ± 1
  An assessment of the condition of the endocrine system on physical examination (normal condition or list of abnormal conditions, if any)
Physical examination results: musculoskeletal system | Screening, day 1, day 8 ± 1, day 15 ± 1, day 22 ± 1, day 29 ± 1
  An assessment of the condition of the musculoskeletal system on physical examination (normal condition or list of abnormal conditions, if any)
Physical examination results: nervous system | Screening, day 1, day 8 ± 1, day 15 ± 1, day 22 ± 1, day 29 ± 1
  An assessment of the condition of the nervous system on physical examination (normal condition or list of abnormal conditions, if any)
Physical examination results: sensory systems | Screening, day 1, day 8 ± 1, day 15 ± 1, day 22 ± 1, day 29 ± 1
  An assessment of the condition of the sensory systems on physical examination (normal condition or list of abnormal conditions, if any)
Physical examination results: skin/visible mucous membranes | Screening, day 1, day 8 ± 1, day 15 ± 1, day 22 ± 1, day 29 ± 1
  An assessment of the condition of the skin/visible mucous membranes on physical examination (normal condition or list of abnormal conditions, if any)
Results of laboratory and instrumental examinations: clinical blood test - hemoglobin | Screening, day 15 ± 1, day 29 ± 1
  Hemoglobin (g/L)
Results of laboratory and instrumental examinations: clinical blood test - hematocrit | Screening, day 15 ± 1, day 29 ± 1
  Hematocrit (%)
Results of laboratory and instrumental examinations: clinical blood test - red blood cell count | Screening, day 15 ± 1, day 29 ± 1
  Red blood cell count (cells/L)
Results of laboratory and instrumental examinations: clinical blood test - platelet count | Screening, day 15 ± 1, day 29 ± 1
  Platelet count (cells/L)
Results of laboratory and instrumental examinations: clinical blood test - leukocyte count | Screening, day 15 ± 1, day 29 ± 1
  Leukocyte count (cells/L)
Results of laboratory and instrumental examinations: clinical blood test - erythrocyte sedimentation rate | Screening, day 15 ± 1, day 29 ± 1
  Erythrocyte sedimentation rate (mm/h)
Results of laboratory and instrumental examinations: clinical blood test - myelocytes | Screening, day 15 ± 1, day 29 ± 1
  Leukocyte formula (myelocytes, %)
Results of laboratory and instrumental examinations: clinical blood test - band neutrophils | Screening, day 15 ± 1, day 29 ± 1
  Leukocyte formula (band neutrophils, %)
Results of laboratory and instrumental examinations: clinical blood test - segmented neutrophils | Screening, day 15 ± 1, day 29 ± 1
  Leukocyte formula (segmented neutrophils, %)
Results of laboratory and instrumental examinations: clinical blood test - eosinophils | Screening, day 15 ± 1, day 29 ± 1
  Leukocyte formula (eosinophils, %)
Results of laboratory and instrumental examinations: clinical blood test - basophils | Screening, day 15 ± 1, day 29 ± 1
  Leukocyte formula (basophils, %)
Results of laboratory and instrumental examinations: clinical blood test - monocytes | Screening, day 15 ± 1, day 29 ± 1
  Leukocyte formula (monocytes, %)
Results of laboratory and instrumental examinations: clinical blood test - lymphocytes | Screening, day 15 ± 1, day 29 ± 1
  Leukocyte formula (lymphocytes, %)
Results of laboratory and instrumental examinations: blood chemistry - glucose | Screening, day 15 ± 1, day 29 ± 1
  Glucose concentration (mmol/L)
Results of laboratory and instrumental examinations: blood chemistry - cholesterol | Screening, day 15 ± 1, day 29 ± 1
  Total cholesterol concentration (mmol/L)
Results of laboratory and instrumental examinations: blood chemistry - protein | Screening, day 15 ± 1, day 29 ± 1
  Total protein concentration (g/L)
Results of laboratory and instrumental examinations: blood chemistry - bilirubin | Screening, day 15 ± 1, day 29 ± 1
  Total bilirubin concentration (micromol/L)
Results of laboratory and instrumental examinations: blood chemistry - creatinine | Screening, day 15 ± 1, day 29 ± 1
  Creatinine concentration (micromol/L)
Results of laboratory and instrumental examinations: blood chemistry - alkaline phosphatase | Screening, day 15 ± 1, day 29 ± 1
  Alkaline phosphatase activity (U/L)
Results of laboratory and instrumental examinations: blood chemistry - alanine transaminase | Screening, day 15 ± 1, day 29 ± 1
  Alanine transaminase activity (U/L)
Results of laboratory and instrumental examinations: blood chemistry - aspartate transaminase | Screening, day 15 ± 1, day 29 ± 1
  Aspartate transaminase activity (U/L)
Results of laboratory and instrumental examinations: blood chemistry - gamma-GTP | Screening, day 15 ± 1, day 29 ± 1
  Gamma-glutaryl transpeptidase activity (U/L)
Results of laboratory and instrumental examinations: urinalysis - specific gravity | Screening, day 15 ± 1, day 29 ± 1
  Specific gravity of the urine
Results of laboratory and instrumental examinations: urinalysis - pH | Screening, day 15 ± 1, day 29 ± 1
  pH of the urine
Results of laboratory and instrumental examinations: urinalysis - protein | Screening, day 15 ± 1, day 29 ± 1
  Protein concentration (g/L)
Results of laboratory and instrumental examinations: urinalysis - glucose | Screening, day 15 ± 1, day 29 ± 1
  Glucose concentration (mmol/L)
Results of laboratory and instrumental examinations: urinalysis - red blood cells | Screening, day 15 ± 1, day 29 ± 1
  Red blood cell content (number in sight)
Results of laboratory and instrumental examinations: urinalysis - white blood cells | Screening, day 15 ± 1, day 29 ± 1
  White blood cell content (number in sight)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - heart rate | Screening, day 1, day 8 ± 1, day 15 ± 1, day 22 ± 1, day 29 ± 1
  12-lead ECG (I, II, III, aVR-enhanced unipolar abduction from the right arm , aVL-enhanced unipolar abduction from the left arm, aVF - enhanced unipolar abduction from the left leg, V1-V6) taken while lying down: heart rate (beats per minute)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - PQ interval | Screening, day 1, day 8 ± 1, day 15 ± 1, day 22 ± 1, day 29 ± 1
  12-lead ECG (I, II, III, aVR-enhanced unipolar abduction from the right arm , aVL-enhanced unipolar abduction from the left arm, aVF - enhanced unipolar abduction from the left leg, V1-V6) taken while lying down: PQ interval (is the period, measured in milliseconds, that extends from the beginning of the P wave (the onset of atrial depolarization) until the beginning of the QRS complex)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - QRS complex | Screening, day 1, day 8 ± 1, day 15 ± 1, day 22 ± 1, day 29 ± 1
  12-lead ECG (I, II, III, aVR-enhanced unipolar abduction from the right arm , aVL-enhanced unipolar abduction from the left arm, aVF - enhanced unipolar abduction from the left leg, V1-V6) taken while lying down: QRS complex (the QRS complex is the combination of three of the graphical deflections seen on a typical electrocardiogram)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - corrected QT interval | Screening, day 1, day 8 ± 1, day 15 ± 1, day 22 ± 1, day 29 ± 1
  12-lead ECG (I, II, III, aVR-enhanced unipolar abduction from the right arm , aVL-enhanced unipolar abduction from the left arm, aVF - enhanced unipolar abduction from the left leg, V1-V6) taken while lying down: corrected QT interval (distance from the beginning of the QRS complex to the end of the T wave) (Frederica correction)

CONTACTS AND LOCATIONS:
Locations (17):
- Russia (17):
  - State autonomous health care institution "Engels City Clinical Hospital No. 1", Engel's
  - Ivanovo Kuvaev Clinical Hospital, Ivanovo
  - State Budgetary Institution of Healthcare of Moscow "City Polyclinic No. 2 of the Moscow Department of Healthcare", Moscow
  - Unimed-C Jsc, Moscow
  - The State Budgetary Healthcare Institution of the Moscow Region "Moscow Regional Research Clinical Institute named after M.F. Vladimirsky", Moscow
  - Limited Liability Company "ErSi Medical", Novosibirsk
  - Professors' Clinic LLC., Perm
  - Limited Liability Company "Medical Center Eco-Safety", Saint Petersburg
  - Limited Liability Company "Energy of Health", Saint Petersburg
  - St. Petersburg State Budgetary Healthcare Institution "City Polyclinic No. 117", Saint Petersburg
  - Limited Liability Company "Clinic Zvezdnaya", Saint Petersburg
  - Limited Liability Company "Meili", Saint Petersburg
  - State Budgetary Institution "St. Petersburg Research Institute of Emergency Care named after I.I. Djanelidze", Saint Petersburg
  - Private institution of higher education "Medical University 'Reavis'", Samara
  - Association "Regional Medical Center 'Open Medicine'", Tolyatti
  - LLC "Polyclinic Polimedika Veliky Novgorod", Veliky Novgorod
  - Limited Liability Company "Medical Center for Diagnosis and Prevention Plus", Yaroslavl

IPD SHARING:
Plan to Share IPD: No